CLINICAL TRIAL: NCT02979067
Title: Improvement of Oxygenation During Apnoea by i-THRIVE (Infant Transnasal Humidified Rapid Insufflation Ventilatory Exchange): A Single-centre Prospective Randomized Controlled Trial.
Brief Title: Improvement of Oxygenation During Apnoea by i-THRIVE
Acronym: i-Thrive
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Insel Gruppe AG, University Hospital Bern (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 2016-01516
Record Dates: First submitted 2016-11-15; First posted 2016-12-01 (Estimated); Last update posted 2017-05-12 (Actual); Status verified 2017-05

CONDITIONS: Preoxygenation
Keywords: Apnoea time, preoxygenation, difficult airway, emergency
MeSH Terms: conditions — Emergencies

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (3):
- High-flow 100% oxygen (Active Comparator): Nasal oxygen flow
  Interventions: Procedure: Nasal oxygen flow
- Low-flow 100% oxygen (Active Comparator): Nasal oxygen flow
  Interventions: Procedure: Nasal oxygen flow
- High-flow 30% oxygen (Active Comparator): Nasal oxygen flow
  Interventions: Procedure: Nasal oxygen flow

INTERVENTIONS:
Procedure: Nasal oxygen flow — Nasal oxygen flow during apnoea

SUMMARY:
Improvement of oxygenation during apnoea by i-THRIVE Infant Transnasal Humidified Rapid Insufflation Ventilatory Exchange A single-centre prospective randomized controlled trial.

DETAILED DESCRIPTION:
High-Flow nasal cannula therapy is the administration of heated, humidified and blended air/oxygen via nasal cannula at rates of at least 2 L/kg bodyweight /min. This high-flow nasal cannula therapy was developed in neonatal intensive care unit for preterm babies with respiratory pauses as an alternative to continuous pressure support (CPAP). Due to its ease of use and safety to apply to a wide range of indication, this oxygen delivery therapy is increasingly gaining interest for providing respiratory support in paediatric and adult patients with respiratory failure in the ICU. High-flow nasal cannula therapy is applied in preterm infant with respiratory distress syndrome, apnoea of prematurity or a respiratory support after extubation. In the adult population the use of HFNCT focuses on hypoxemic respiratory failure and improvement reduction of hypoxemia during intubation in the anesthesia environment. A new application for high-flow nasal cannula therapy in adults is the extension of apnoea time in patients with difficult airways who are undergoing general anesthesia. In this environment a new term for this kind of oxygen therapy was created: THRIVE transnasal humidified rapid-insufflation ventilatory exchange. To distinguish this kind of high-flow nasal cannula therapy in apnoeic patients from the one in the paediatric ICU or ward the investigators use the term i-THRIVE for infant transnasal humidified rapid insufflation ventilation exchange.

Due to the increased oxygen consumption and the reduced functional residual capacity, neonates, infants, and small children have a reduced apnoea tolerance compared to adults. Furthermore infants and small children have a greater closing capacity, which increases the airway collapse under general anesthesia and muscle paralysis. A direct consequence is that hypoxemia is very likely to occur after cessation of spontaneous or assisted ventilation during induction of anesthesia. Apnoea without supplemental oxygen leads to hypoxemia in a 1-year-old infant without preoxygenation within seconds. All paediatric (and adult) patients undergoing general anesthesia have at least a brief period of apnoea during intubation between the time the face-mask is removed from the patient and the tube is placed in the trachea. Therefore, at least short phases of deoxygenation may occur.

However if anesthesia needs to be provided in emergency situations or in the presence of a difficult airway, the rate of complication increases rapidly. In these circumstances methods that reduce desaturation incidents during prolonged difficult intubation are desirable. Due to oxygen toxicity in neonates or small children, prevention of hypoxemia with oxygen concentration below 60% would be favourable in this setting. Despite promising pilot results with high-flow nasal cannula therapy, it is unknown whether this technique is superior to low-flow oxygenation with high concentration and whether it is necessary to apply high-flow nasal cannula therapy with high (80-100%) versus low (30-50%) concentration oxygen.

This study investigates under controlled circumstances the concept of i-THRIVE to prolong the apnoea time without deoxygenation and to improve safety of airway management in paediatric patients. Furthermore, this study enables to quantify the effects of different oxygen concentrations with high-flow nasal cannula therapy and distinguishes it better from conventional low-flow apnoeic oxygenation methods.

ELIGIBILITY:
Inclusion Criteria:

* 10-20 kg
* ASA 1+2
* Written informed consent
* Speaking German

Exclusion Criteria:

* Difficult intubation
* Oxygen dependency
* Congenital heart or lung disease
* BMI >30g/m2
* High aspiration risk
* nasal obstruction

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2016-12 (Actual); Primary Completion 2017-05 (Actual); Study Completion 2017-05 (Actual)

PRIMARY OUTCOMES:
Time until desaturation from SpO2 100% to 95% measured by pulse oxymetry | up to ten minutes during intervention

SECONDARY OUTCOMES:
TcCO2mmHg level | study intervention, around 15 minutes
TcO2mmHg level | study intervention, around 15 minutes

CONTACTS AND LOCATIONS:
Overall Officials: Robert Greif, MD MME FERC, Study Chair — University hospital Bern and University of Bern
Locations (1):
- Bern University Hospital and University of Bern, Bern, Switzerland

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Riva T, Pedersen TH, Seiler S, Kasper N, Theiler L, Greif R, Kleine-Brueggeney M. Transnasal humidified rapid insufflation ventilatory exchange for oxygenation of children during apnoea: a prospective randomised controlled trial. Br J Anaesth. 2018 Mar;120(3):592-599. doi: 10.1016/j.bja.2017.12.017. Epub 2018 Jan 27. PMID 29452816